CLINICAL TRIAL: NCT01971203
Title: Double-blind, Randomized, Active Controlled Study of the Efficacy and Safety of Extended-release Quetiapine Fumarate (Seroquel XR) as Adjunctive Medication Therapy to Cognitive Behavioral Therapy in the Treat,Ent of Patients With Comorbid Major Depression and Generalized Anxiety Disorder
Brief Title: Efficacy of Extended-release Quetiapine (Seroquel XR) as Adjunctive Therapy to Cognitive Behavioral Therapy in the Treat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Jack Hirschowitz, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 09-0807
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Major Depressive Disorder; Generalized Anxiety Disorder
Keywords: seroquel XR; quetiapine XR; major depression; generalized anxiety disorder; CBT; co-morbid MDD
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- seroquel xr (Experimental): quetiapine target dosage will be 150 mg/day, beginning at 50 mg/day 16 weeks of treatment including CBT
  Interventions: Drug: seroquel xr
- placebo plus CBT (Placebo Comparator): treatment group receiving placebo pill plus CBT
  Interventions: Behavioral: CBT

INTERVENTIONS:
Drug: seroquel xr — Quetiapine target dosage will be 150 mg/day, beginning at 50 mg/day
  Other Names: quetiapine XR
  Arms: seroquel xr
Behavioral: CBT — 16 weeks of treatment
  Other Names: cognitive behavioral therapy
  Arms: placebo plus CBT

SUMMARY:
The primary objective of the study is to determine whether quetiapine extended-release in combination with cognitive behavioral therapy (CBT) is more effective than CBT plus placebo in treating depressive and anxiety symptoms in patients with both major depression and generalized anxiety disorder. Approximately 64 individuals (adults 18-65) will be randomly assigned to treatment group for 16 weeks. Weekly CBT sessions will be conducted lasting about 45 minutes and weekly visits with the study psychiatrist lasting about 20 minutes in which medication will be discussed. Both clinician administered and self-report measures will be used to compare groups before and after 16 weeks.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of quetiapine extended-release as adjunctive therapy to cognitive behavioral therapy (CBT) compared to CBT plus placebo in the treatment of patients with comorbid major depression and generalized anxiety disorder. We will also evaluate the quality of life in patients with comorbid MDD/GAD, the response and remission rates by treatment group, changes in sleep quality, and tolerability of adjunctive quetiapine to CBT.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* A diagnosis of both major depression (single episode or recurrent) and generalized anxiety disorder by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
* Females and/or males aged 18 to 65 years
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrollment
* Able to understand and comply with the requirements of the study

Exclusion Criteria:

* Pregnancy or lactation
* Any history of psychosis, bipolar disorder, schizophrenia, eating disorders or OCD
* Imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrollment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomization
* Substance or alcohol dependence at enrollment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* Substance abuse by DSM-IV criteria within 6 months prior to enrollment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrollment or randomization of treatment in the present study
* Participation in another drug trial within 4 weeks prior to enrollment into this study or longer in accordance with local requirements
* A patient with Diabetes Mellitus (DM)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Hirschowitz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the Mount Sinai faculty referrals, medical center employee newsletter, and advertisements in local newspapers, radio, and craigslist.
Pre-assignment Details: Ninety-four participants were screened - 10 participants did not meet study eligibility, 22 elected not to continue. 62 participants were randomized, but 7 never returned for the first visit, leaving 55 participants who began treatment.
Groups:
- Seroquel XR Plus CBT: Participants were required to take a minimum of one 50 mg pill of quetiapine XR a day with an intended titration schedule reaching 150 mg over the first three weeks, adding one pill per week. . If a participant could not tolerate the increased dose, then dosage was decreased to either one or two pills a day.
  All participants who completed the study received 16 sessions of CBT and discontinued medication at 16 weeks. Although conducted weekly, CBT and medication schedules did not always terminate at the same time.
- Placebo Plus CBT: matching placebo pills plus 16 weeks of Cognitive Behavioral Therapy
Period: Overall Study
Arm/Group | Seroquel XR Plus CBT | Placebo Plus CBT
Started | 26 | 29
Completed | 17 | 21
Not Completed | 9 | 8
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seroquel XR Plus CBT | Placebo Plus CBT | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.93 (13.68) | 39.88 (12.81) | 39.90 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 13 | 11 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 22 | 41
  Black | 4 | 4 | 8
  Hispanic | 2 | 3 | 5
  Asian | 3 | 1 | 4
  Other | 2 | 1 | 3
  Unknown | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  Less than HS | 1 | 0 | 1
  HS | 4 | 2 | 6
  Part college | 3 | 10 | 13
  College | 13 | 15 | 28
  Advanced | 8 | 4 | 12
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Secondary Outcome: HAM-A
Description: Hamilton Rating Scale for Anxiety (HAM-A) is a 14-item clinician-administered scale measuring symptoms with total scale from 0 (not present) to 56 (severe) to severe anxiety.
Time Frame: baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Seroquel XR Plus CBT: Participants were required to take a minimum of one 50 mg pill of quetiapine XR a day.
Arm/Group | Seroquel XR Plus CBT | Placebo Plus CBT
Number analyzed (Participants) | 26 | 29
units on a scale
  Baseline | 16.7 (5.2) | 17.8 (4.7)
  LOCF (last observation carried forward) | 5.9 (3.9) | 9.4 (7.7)

2. Secondary Outcome: Clinical Global Impression Scales for Severity and Improvement
Description: The Clinical Global Impression Scales for Severity and Improvement (CGI-I and CGI-S), both clinician rated, measures overall severity of symptoms and level of improvement on a seven-point scale from 0 (not applicable or not assessed) to 7, where 7 is the most severe. In order for a participant to be considered a treatment responder, he or she must receive a score of 1 (not ill or very much improved) or 2 (borderline mentally ill or much improved).
Time Frame: up to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR Plus CBT | Placebo Plus CBT
Number analyzed (Participants) | 26 | 29
units on a scale
  CGI-S Baseline | 4.1 (0.5) | 4.3 (0.5)
  CGI-S LOCF | 2.5 (1.2) | 2.9 (1.2)
  CGI-I Baseline | 3.3 (1.6) | 2.7 (1.9)
  CGI-I LOCF | 1.8 (1.0) | 2.4 (1.1)

3. Secondary Outcome: Changes in Sexual Functioning Questionnaire (CSFQ)
Description: Changes in Sexual Functioning Questionnaire (CSFQ) at week 16 as compared to baseline. The CSFQ assesses interest, functioning, and satisfaction in sex on a six-point scale, where 1 is greater than normal and 6 is totally absent, with full range from 5 (greater than normal) to 30 (totally absent).
Time Frame: baseline and week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR Plus CBT | Placebo Plus CBT
Number analyzed (Participants) | 26 | 29
units on a scale
  Baseline | 15.1 (6.3) | 16.6 (5.7)
  LOCF | 1.8 (0.9) | 14.1 (6.5)

4. Primary Outcome: MADRS
Description: Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician-administered, with overall score ranges from 0 (normal) to 54 (severe depression). Score at 16 weeks as compared to baseline.
Time Frame: baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR Plus CBT | Placebo Plus CBT
Number analyzed (Participants) | 26 | 29
units on a scale
  Baseline | 27.1 (5.5) | 28.6 (6.5)
  LOCF (last observation carried forward) | 9.1 (6.9) | 15.7 (11.9)

ADVERSE EVENTS:
Arm/Group | Seroquel XR Plus CBT | Placebo Plus CBT
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29
Other Adverse Events (participants affected / at risk) | 24/26 | 11/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seroquel XR Plus CBT (N=26) | Placebo Plus CBT (N=29)
depression (Psychiatric disorders) | 1 | 0
Blood clot (Blood and lymphatic system disorders) | 1 | 0
Sedation (Nervous system disorders) | 24 | 11

LIMITATIONS AND CAVEATS:
The limitations of this research are the small sample size and the high rate of subject drop-out between randomization and initiation of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes